CLINICAL TRIAL: NCT01866280
Title: Effect of Sleep Timing, Independent of Duration, on Food Intake and Metabolic Control of Energy Balance
Brief Title: Sleep Timing and Energy Balance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Luke's-Roosevelt Hospital Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: ST-01
Record Dates: First submitted 2013-04-24; First posted 2013-05-31 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2015-04

CONDITIONS: Sleep; Meals
Keywords: Sleep; Sleep duration; Meals; Food intake; Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Normal sleep Normal meals (Experimental): Normal sleep/Normal meal times
  Interventions: Behavioral: Normal sleep; Behavioral: Normal meals
- Normal sleep Late meals (Experimental): Normal sleep/Late meal times
  Interventions: Behavioral: Normal sleep; Behavioral: Late meals
- Late sleep Late meals (Experimental): Late sleep/Late meal times
  Interventions: Behavioral: Late sleep; Behavioral: Late meals
- Late sleep Normal meals (Experimental): Late sleep/Normal meal times
  Interventions: Behavioral: Normal meals; Behavioral: Late sleep

INTERVENTIONS:
Behavioral: Normal sleep — Normal sleep= sleep 2300-0700
  Arms: Normal sleep Late meals; Normal sleep Normal meals
Behavioral: Normal meals — Normal meal times=approximately 1.5, 5, and 11 h after wake up for breakfast, lunch, and dinner, and snack at 13 h after wake up time
  Arms: Late sleep Normal meals; Normal sleep Normal meals
Behavioral: Late sleep — Late sleep=sleep at 0230-1030 hours
  Arms: Late sleep Late meals; Late sleep Normal meals
Behavioral: Late meals — Late meal times= approximately 4.5, 7, and 13 h after wake up time for breakfast, lunch and dinner, and snack at 15 h.
  Arms: Late sleep Late meals; Normal sleep Late meals

SUMMARY:
The purpose of this study is to test the effects of sleep and meal timing, independent of sleep duration, on glucose regulation and metabolic and hormonal control of energy balance in normal weight adults.

This study will be a 4-phase, randomized controlled study of 5 days each in which participants will undergo 2 phases of late sleep times that differ in meal timing (normal or late) and 2 phases of normal sleep times that differ in meal timing (normal or late).

The Aims and Hypotheses of this study are:

Aim 1: To compare hormonal regulation of food intake and metabolic risk markers in response to altered sleep and meal timing.

* Hypothesis 1: There will be an interaction between sleep and meal time on glucose, insulin, and glucose and insulin area under the curve after the glucose tolerance test such that the late sleep/late meal will result in the worst metabolic profile, normal sleep/late meal and late sleep/normal meal will have an intermediate profile, and normal sleep/normal meal will result in the best metabolic profile.
* Hypothesis 2: There will be an interaction between sleep and meal time on leptin and ghrelin concentrations such that the late sleep/late meal timing phase will result in low leptin/high ghrelin, normal sleep/late meal timing and late sleep/normal meal will have an intermediate profile, and normal sleep/normal meal timing will result in high leptin/low ghrelin.

Aim 2: To compare food intake over a 24-h period in response to altered sleep and meal timing.

• Hypothesis 3: Energy and fat intakes will be greater during the late sleep timing phase compared to normal sleep timing.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index 22-25
* Normal scores on sleep questionnaires (PSQI, ESS, Berlin, SDIQ)
* Normal score on Beck Depression Inventory
* Intermediate chronotype on Composite Scale of Morningness/Eveningness

Exclusion Criteria:

* Neurological, medical, or psychiatric disorders
* Eating disorders
* Diabetes
* Sleep disorders
* Travel across time zones
* History of drug/alcohol abuse
* Caffeine intake >300 mg/d
* Excessive daytime sleepiness
* Pregnancy or within 1 y post-partum

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2012-11; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Food intake | Single day
  Ad libitum food intake will be assessed on day 5
Oral Glucose Tolerance | 2 hours
  Oral glucose tolerance test will be performed at scheduled breakfast time on day 4
Meal tolerance test | 3 hours
  Glucose and insulin responses to a liquid meal will be assessed at scheduled lunch time

SECONDARY OUTCOMES:
Hormonal profile | 24 hours
  On day 3, the following hormones will be assessed from overnight hours: glucose, insulin, cortisol, melatonin, leptin, ghrelin, PYY, GLP-1

CONTACTS AND LOCATIONS:
Locations (1):
- St. Luke's/Roosevelt Hospital, New York, New York, United States